CLINICAL TRIAL: NCT06981728
Title: Ultrasound-Guided Mid-Point Transverse Process to Pleura Block Versus Thoracic Paravertebral Block for Pain Management in Patients With Multiple Rib Fractures (A Prospective Randomized Double- Blinded, Non-inferiority Trial )
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Yassien Mahmoud Ahmed, MD doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: fracture ribs
Record Dates: First submitted 2025-05-12; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: According to computer-generated software randomization (www.randomization.com) table into two groups of 35 each, patients randomly were allocated to Group M or Group P at a ratio of 1:1.
  * Group M: mid-point transverse to pleura block.
  * Group P: thoracic paravertebral block. The grouping sequence was put into a sealed opaque envelope, the operator opened the envelope to identify the type of block. Patients were blinded to the grouping assignments. After trial completion, all participants remained unaware of the grouping assignments until un blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M (MTPB) (Active Comparator): Mid-point transverse to pleura block
  Interventions: Procedure: Mid point transverse to pleura block
- P (TPVB) (Sham Comparator): Thoracic paravertebral block
  Interventions: Procedure: Mid point transverse to pleura block

INTERVENTIONS:
Procedure: Mid point transverse to pleura block — TPVB and MTPB was performed at a spinal level midway between the uppermost and the lowest fractured rib, with the patient in a sitting position, and under complete aseptic conditions, a linear ultrasound probe (GE Healthcare-Logiq F6) will be placed oblique parasagittally 3 cm lateral to spinous process used to identify the transverse process, pleura, superior costotransverse ligament, and the paravertebral space at the target vertebral level.
  After skin and subcutaneous tissue infiltration with 2-3 mL of 2% lignocaine, an 18-gauge Touhy needle was inserted under ultrasound guidance until the needle tip reaches :
  * the midpoint between the transverse process and the pleura (group M).
  * the paravertebral space (group P). A bolus dose (0.3mL/kg) of plain bupivacaine 0.5% plus 8 mg of dexamethasone was injected after negative aspiration to blood and air.
  Other Names: Thoracic paravertebral block

SUMMARY:
The aim of our study is to investigate whether the analgesic effect of MTPB is non inferior to that of TPVB in trauma patients with multiple rib fractures.

DETAILED DESCRIPTION:
Trauma is a major global health problem. In Egypt, trauma-related death accounted for 8% of total fatalities and was the eighth leading cause of death in 2010. However.[1]Rib fractures have an incidence around 10% of all trauma patients and over 30% of chest trauma patients.[2] Multiple fractured ribs are associated with extreme pain, to avoid intensifying discomfort, patients' breathing becomes shallower and they repress coughing, leading to respiratory insufficiency. Which may result in numerous complications, as sputum retention, atelectasis, infection, and respiratory insufficiency. This is associated with increase in intensive care admissions and mortality (25%).[3] Hence, pain control is the cornerstone of rib fracture management. Modalities for pain relief ranges from oral administration of analgesic drugs to regional nerve blocks including [intrapleural, intercostal ,thoracic paravertebral nerve blockade (TPVB)]. Despite the low rate of technical failure in TPVB execution (6.1%), pulmonary complications, such as inadvertent pleural puncture (0.8%) and pneumothorax (0.5%), are still a recognized risk.[4] Bedside ED-performed ultrasound-guided anesthesia is gaining in popularity, and early and adequate pain control has shown improved patient outcomes with rare complications.

One of the most recently described technique is mid-point transverse process to pleura (MTP) block.[2] In MTP block, the local anesthetic drug is deposited at the mid-point between the transverse process and pleura and it reaches the paravertebral space by diffusion. With this technique, even if superior costotransverse ligament (SCTL) is not visible, effective block can be achieved. In addition, needle is placed far away from pleura minimizing the rate of pneumothorax.[5]

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 18 and 70 years, from both genders, who had uni lateral traumatic multiple rib fractures (three or more confirmed by a CT chest scan).

Exclusion Criteria:

* Significant head injury/unconsciousness (GCS less than 15).
* Patients with Pain score >6.
* those having significant trauma outside the chest wall, e.g., acute spine or pelvic fracture, severe traumatic brain or spinal cord injury, or abdominal visceral injuries.
* Obese patients with body mass index ≥ 35.
* coagulopathy.
* History of drug allergy to local anesthetics.
* Patient refusal.
* Local infection at the injection site.
* Opioid addiction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the mean difference in numeric rating pain scores (NRS) between the MTPB and TPVB groups at 24-hour after the block. | 24hour

SECONDARY OUTCOMES:
• NRS scores at different times up to 24 hours. | 72hour
Time for first analgesic request. • Total 24 hours analgesic consumption. | 24hour
• Total 24 hours analgesic consumption. | 24hour
• Time for block performance. | 30min
• Dermatomal block effect. | 24hour
inspiratory volumes (mL) measured with a volume incentive spirometer. | 72hour
respiratory rate (RR),Heart rate (HR), Blood Pressure (BP), peripheral oxygen saturation (SpO2),and need for mechanical ventilation. | 3 days
• Complications such as pneumothorax bradycardia hypotension. • development of pneumonia, hospital length of stay, and mortality. | 3days

CONTACTS AND LOCATIONS:
Overall Officials: alaa attia, professor, Study Director — alaaguhina@aun.edu.eg; Monira Ismail, professor, Study Director — Monira.taha77@med.suez.edu.eg; muhamed mamdouh, lecturer, Study Director — mamdouh372@med.aun.edu.eg

REFERENCES:
- See also: Related Info — https://goo.gl/MTv7ea
- See also: Related Info — https://goo.gl/AeNXBz